CLINICAL TRIAL: NCT00892047
Title: Incomplete Response in Late Life Depression: Getting to Remission
Brief Title: Incomplete Response in Late Life Depression: Getting to Remission (IRL GREY)
Acronym: IRL GREY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Charles Reynolds, Director NIMH Center of Excellence in the Prevention and Treatment of Depression in Older Adults; UPMC Endowed Professor in Geriatric Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MH083660-01A1
Record Dates: First submitted 2009-04-29; First posted 2009-05-04 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Depression
Keywords: Depression; Aripiprazole; Venlafaxine; Partial Remission; Augmentation strategy; Treatment resistance; Elderly; Late-life
MeSH Terms: conditions — Depression | interventions — Aripiprazole; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: venlafaxine plus aripiprazole (Experimental): antidepressant (venlafaxine) plus aripiprazol or venlafaxine plus placebo
  Interventions: Drug: venlafaxine XR plus aripiprazole
- 2: Placebo Comparator (Experimental): antidepressant (venlafaxine) plus aripiprazol or venlafaxine plus placebo
  Interventions: Drug: venlafaxine plus placebo

INTERVENTIONS:
Drug: venlafaxine XR plus aripiprazole — Dosage varies. Subject remains on antidepressant throughout the 36 week study. Will be randomized to aripiprazole or placebo for up to 24 weeks.
  Other Names: effexor XR, abilify
  Arms: 1: venlafaxine plus aripiprazole
Drug: venlafaxine plus placebo — Dosage varies. Subject remains on antidepressant throughout the 36 week study. Will be randomized to aripiprazole or placebo for up to 24 weeks.
  Arms: 2: Placebo Comparator

SUMMARY:
The primary aims of this study are to:

1. Assess the efficacy of aripiprazole augmentation for the acute and continuation treatment of TRLLD.

   Hypothesis 1: Patients with TRLLD (defined as those who do not remit after 12 weeks of acute treatment with venlafaxine XR) will have a higher rate of remission with aripiprazole than with placebo augmentation (primary outcome) and greater improvement in depressive symptoms and stability of remission (secondary outcomes).
2. Assess the tolerability of aripiprazole in TRLLD with a focus on adiposity and akathisia/restlessness.

Hypothesis 2: Aripiprazole will be associated with a higher rate of clinically significant akathisia and increased adiposity than placebo.

The Secondary/exploratory aims of this study are to:

1. Examine anxiety, medical burden, and executive impairment as moderators of aripiprazole augmentation efficacy in TRLLD.

   Hypothesis 3: Pre-levels of anxiety symptoms, medical burden, and executive impairment will be treatment-specific factors: they will moderate the efficacy of aripiprazole augmentation. The aripiprazole-placebo difference will be greater in individuals with these variables, compared to those without these variables because these three factors will be associated with a decreased likelihood that "staying the course" with venlafaxine monotherapy will achieve remission.
2. Examine genetic predictors (phase 1) and moderators (phase 2-3) of treatment outcomes, while controlling for drug exposure.

Hypothesis 4: Selected polymorphisms will reduce remission rate with venlafaxine and will reduce efficacy and tolerability with aripiprazole.

DETAILED DESCRIPTION:
Incomplete response in the treatment of late-life depression (LLD) is a large public health challenge: at least 50% of older people fail to respond adequately to antidepressant pharmacotherapy, even under optimal treatment conditions. Treatment resistant late-life depression (TRLLD) increases risk for early relapse, undermines adherence to treatment for coexisting medical disorders, amplifies disability and cognitive impairment, imposes greater burden on family caregivers, and increases the risk for early mortality, including suicide. Getting to and sustaining remission is the primary goal of treatment, yet there is a paucity of controlled studies of how best to manage TRLLD.

This is a multi-site study being conducted by 3 sites: University of Pittsburgh, University of Toronto, and Washington University. We propose to enroll 500 subjects aged 60 and older with major depressive disorder at this site and treat them openly for 12 weeks with venlafaxine XR (up to 300mg/d) (phase 1). Participants meeting criteria for incomplete response will be randomly assigned to receive either aripiprazole (2-15 mg/d; target dose: 10 mg/d) or placebo augmentation (adding a pill without active medicine) of venlafaxine for 12 weeks (phase 2), with the goal of achieving remission (MADRS≤10 for two consecutive assessments). Those who remit in phase 2 will receive continuation treatment, with the same double-blinded intervention to which they were randomly assigned (phase 3), for 12 weeks to determine the stability of remission. Efficacy and tolerability data will provide a clinically informative estimate of benefits and risks of aripiprazole augmentation for TRLLD.

In addition to the primary goal of assessing these benefits and risks, we will develop evidence relevant to personalized treatment for LLD by testing the roles of clinical (comorbid anxiety, medical burden, and executive impairment) and genetic (selected polymorphisms in serotonin, norepinephrine, and dopamine genes) variables, while controlling for variability in drug exposure for efficacy and tolerability analyses. This approach will allow us to distinguish treatment-specific resistance factors versus general prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 60 years.
2. Major depressive disorder (MDD), single or recurrent, as diagnosed by the SCID-IV.
3. MADRS ≥ 15.

Exclusion Criteria:

1. Inability to provide informed consent.
2. Depressive symptoms not severe enough (i.e., MADRS < 15) at the baseline assessments.
3. Dementia based upon DSM-IV criteria as well as a Folstein MMSE score of less than 24. Patients screened out due to dementia will be referred to a memory clinic or to the UPMC Alzheimer's Disease Research Center for evaluation to clarify the presence or absence of a dementia.
4. Lifetime diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms, as diagnosed by the SCID. A recommendation for psychiatric referral will be made in these cases.
5. Abuse of or dependence on alcohol or other substances within the past 3 months as determined by SCID, and confirmed by study physician interview.
6. High risk for suicide (e.g., active SI and/or current/recent intent or plan) AND unable to be managed safely in the clinical trial (e.g., unwilling to be hospitalized). Urgent psychiatric referral will be made in these cases.
7. Contraindication to venlafaxine XR or aripiprazole as determined by study physician including history of intolerance of either venlafaxine XR or aripiprazole in the study target dosage range (venlafaxine XR at up to 225 mg/day; aripiprazole at up to 15mg/day).
8. Failure to respond to at least 6 weeks of venlafaxine (>225 mg/d) plus aripiprazole (>10 mg/d).
9. Inability to communicate in English (i.e., interview cannot be conducted without an interpreter; subject largely unable to understand questions and cannot respond in English).
10. Non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview)
11. Unstable medical illness, including delirium, uncontrolled diabetes mellitus, hypertension, hyperlipidemia, or cerebrovascular or cardiovascular risk factors that are not under medical management. This will be determined based on information from the patient's personal physician's and study physician clinical judgment. Referral to the patient's personal physician or to a general practitioner will be made in these cases.
12. Subjects taking psychotropic medications that cannot be safely tapered or discontinued prior to study initiation: this would include patients on Monoamine Oxidase Inhibitors (MAOI) who would need to be off the MAOI for 14 days to be eligible for the study to avoid adverse drug interactions. Patients will not be allowed to take antidepressant or atypical antipsychotic medication other than the study medication, unless it is a low dose antidepressant prescribed for chronic pain that would not be medically advisable to stop (e.g., amitryptyline 50mg). If a patient's depression is adequately treated on his/her psychotropic medication, he/she would not be eligible for the study. If a patient failed a trial of venlafaxine (12 weeks of treatment with venlafaxine including at least 6 weeks on 300mg/day), he/she would not be eligible. The following are allowed: benzodiazepines up to 2mg/d lorazepam equivalent; other sedative-hypnotics (e.g., zolpidem, zaleplon, eszopiclone); gabapentin if prescribed for non-psychiatric indication (e.g., neuropathy). Except for MAOIs, there is really no clinical rationale to exclude patients on specific concomitant medications unless they are medically unstable (in which case they are excluded from participation). As noted, patients on an MAOI would need to be off the MAOI for 14 days to protect from adverse drug interactions.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2009-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles F. Reynolds, MD, Principal Investigator — University of Pittsburgh; Eric Lenze, MD, Principal Investigator — Washington University School of Medicine, St. Louis; Benoit Mulsant, MD, Principal Investigator — University of Toronto
Locations (3):
- United States (2):
  - Washington University School of Medicine, St. Louis, St Louis, Missouri
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Result] Lenze EJ, Mulsant BH, Blumberger DM, Karp JF, Newcomer JW, Anderson SJ, Dew MA, Butters MA, Stack JA, Begley AE, Reynolds CF 3rd. Efficacy, safety, and tolerability of augmentation pharmacotherapy with aripiprazole for treatment-resistant depression in late life: a randomised, double-blind, placebo-controlled trial. Lancet. 2015 Dec 12;386(10011):2404-12. doi: 10.1016/S0140-6736(15)00308-6. Epub 2015 Sep 27. PMID 26423182
- [Derived] Olgiati P, Fanelli G, Serretti A. Age or age of onset: which is the best criterion to classify late-life depression? Int Clin Psychopharmacol. 2023 Jul 1;38(4):223-230. doi: 10.1097/YIC.0000000000000472. Epub 2023 Mar 21. PMID 36961017
- [Derived] Ainsworth NJ, Brender R, Gotlieb N, Zhao H, Blumberger DM, Karp JF, Lenze EJ, Nicol GE, Reynolds CF, Wang W, Mulsant BH. Association between lean muscle mass and treatment-resistant late-life depression in the IRL-GRey randomized controlled trial. Int Psychogeriatr. 2023 Dec;35(12):707-716. doi: 10.1017/S1041610222000862. Epub 2023 Jan 3. PMID 36594430
- [Derived] Diniz BS, Mulsant BH, Reynolds CF 3rd, Blumberger DM, Karp JF, Butters MA, Mendes-Silva AP, Vieira EL, Tseng G, Lenze EJ. Association of Molecular Senescence Markers in Late-Life Depression With Clinical Characteristics and Treatment Outcome. JAMA Netw Open. 2022 Jun 1;5(6):e2219678. doi: 10.1001/jamanetworkopen.2022.19678. PMID 35771573
- [Derived] Altmann H, Stahl ST, Gebara MA, Lenze EJ, Mulsant BH, Blumberger DM, Reynolds CF 3rd, Karp JF. Coprescribed Benzodiazepines in Older Adults Receiving Antidepressants for Anxiety and Depressive Disorders: Association With Treatment Outcomes. J Clin Psychiatry. 2020 Sep 29;81(6):20m13283. doi: 10.4088/JCP.20m13283. PMID 32991792
- [Derived] Buchalter ELF, Oughli HA, Lenze EJ, Dixon D, Miller JP, Blumberger DM, Karp JF, Reynolds CF 3rd, Mulsant BH. Predicting Remission in Late-Life Major Depression: A Clinical Algorithm Based Upon Past Treatment History. J Clin Psychiatry. 2019 Dec 10;80(6):18m12483. doi: 10.4088/JCP.18m12483. PMID 31846575
- [Derived] Wei W, Karim HT, Lin C, Mizuno A, Andreescu C, Karp JF, Reynolds CF 3rd, Aizenstein HJ. Trajectories in Cerebral Blood Flow Following Antidepressant Treatment in Late-Life Depression: Support for the Vascular Depression Hypothesis. J Clin Psychiatry. 2018 Oct 23;79(6):18m12106. doi: 10.4088/JCP.18m12106. PMID 30358242
- [Derived] Hsu JH, Mulsant BH, Lenze EJ, Sanches M, Karp JF, Reynolds CF, Blumberger DM. Clinical Predictors of Extrapyramidal Symptoms Associated With Aripiprazole Augmentation for the Treatment of Late-Life Depression in a Randomized Controlled Trial. J Clin Psychiatry. 2018 Jun 19;79(4):17m11764. doi: 10.4088/JCP.17m11764. PMID 29924506
- [Derived] Cristancho P, Lenze EJ, Dixon D, Miller JP, Mulsant BH, Reynolds CF 3rd, Butters MA. Executive Function Predicts Antidepressant Treatment Noncompletion in Late-Life Depression. J Clin Psychiatry. 2018 May/Jun;79(3):16m11371. doi: 10.4088/JCP.16m11371. PMID 29659205
- [Derived] Marshe VS, Maciukiewicz M, Rej S, Tiwari AK, Sibille E, Blumberger DM, Karp JF, Lenze EJ, Reynolds CF 3rd, Kennedy JL, Mulsant BH, Muller DJ. Norepinephrine Transporter Gene Variants and Remission From Depression With Venlafaxine Treatment in Older Adults. Am J Psychiatry. 2017 May 1;174(5):468-475. doi: 10.1176/appi.ajp.2016.16050617. Epub 2017 Jan 10. PMID 28068779
- [Derived] Smagula SF, Karim HT, Lenze EJ, Butters MA, Wu GF, Mulsant BH, Reynolds CF, Aizenstein HJ. Gray matter regions statistically mediating the cross-sectional association of eotaxin and set-shifting among older adults with major depressive disorder. Int J Geriatr Psychiatry. 2017 Dec;32(12):1226-1232. doi: 10.1002/gps.4585. Epub 2016 Sep 19. PMID 27645461
- [Derived] Smagula SF, Lotrich FE, Aizenstein HJ, Diniz BS, Krystek J, Wu GF, Mulsant BH, Butters MA, Reynolds CF 3rd, Lenze EJ. Immunological biomarkers associated with brain structure and executive function in late-life depression: exploratory pilot study. Int J Geriatr Psychiatry. 2017 Jun;32(6):692-699. doi: 10.1002/gps.4512. Epub 2016 Jun 10. PMID 27282141
- [Derived] Kaneriya SH, Robbins-Welty GA, Smagula SF, Karp JF, Butters MA, Lenze EJ, Mulsant BH, Blumberger D, Anderson SJ, Dew MA, Lotrich F, Aizenstein HJ, Diniz BS, Reynolds CF 3rd. Predictors and Moderators of Remission With Aripiprazole Augmentation in Treatment-Resistant Late-Life Depression: An Analysis of the IRL-GRey Randomized Clinical Trial. JAMA Psychiatry. 2016 Apr;73(4):329-36. doi: 10.1001/jamapsychiatry.2015.3447. PMID 26963689
- [Derived] Kasckow J, Youk A, Anderson SJ, Dew MA, Butters MA, Marron MM, Begley AE, Szanto K, Dombrovski AY, Mulsant BH, Lenze EJ, Reynolds CF 3rd. Trajectories of suicidal ideation in depressed older adults undergoing antidepressant treatment. J Psychiatr Res. 2016 Feb;73:96-101. doi: 10.1016/j.jpsychires.2015.11.004. Epub 2015 Nov 19. PMID 26708830
- [Derived] Smagula SF, Butters MA, Anderson SJ, Lenze EJ, Dew MA, Mulsant BH, Lotrich FE, Aizenstein H, Reynolds CF 3rd. Antidepressant Response Trajectories and Associated Clinical Prognostic Factors Among Older Adults. JAMA Psychiatry. 2015 Oct;72(10):1021-8. doi: 10.1001/jamapsychiatry.2015.1324. PMID 26288246
- [Derived] Hall CA, Simon KM, Lenze EJ, Dew MA, Begley A, Butters MA, Blumberger DM, Stack JA, Mulsant B, Reynolds CF 3rd. Depression Remission Rates Among Older Black and White Adults: Analyses From the IRL-GREY Trial. Psychiatr Serv. 2015 Dec 1;66(12):1303-11. doi: 10.1176/appi.ps.201400480. Epub 2015 Aug 17. PMID 26278231
- [Derived] Joel I, Begley AE, Mulsant BH, Lenze EJ, Mazumdar S, Dew MA, Blumberger D, Butters M, Reynolds CF 3rd; IRL GREY Investigative Team. Dynamic prediction of treatment response in late-life depression. Am J Geriatr Psychiatry. 2014 Feb;22(2):167-76. doi: 10.1016/j.jagp.2012.07.002. Epub 2013 Feb 6. PMID 23567441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 3 Centers (University of Pittsburgh, Centre for Addiction and Mental Health in Toronto, Canada, and Washington University). The first participant was enrolled July 2009, last finished August 2014.
Pre-assignment Details: 468 signed consent. 181 were randomized. Of these 181, 91 randomized to venlafaxine plus aripirazol and 90 to venlafaxine plus placebo. Prior to randomization, 191 responded to venlafaxine; 40 withdrew consent; 41 withdrawn by PI, possible AE, 14 non-compliance; 1 death.
Groups:
- 1: Venlafaxine Plus Aripiprazole: antidepressant (venlafaxine) plus aripiprazol or venlafaxine plus placebo
  venlafaxine XR plus aripiprazole: Dosage varies. Subject remains on antidepressant throughout the 36 week study and also receives aripiprazole 2mg to 15mg daily for up to 24 weeks.
- 2: Placebo Comparator: antidepressant (venlafaxine) plus aripiprazol or venlafaxine plus placebo
  venlafaxine plus placebo: Dosage varies. Subject remains on antidepressant throughout the 36 week study and also receives placebo for up to 24 weeks.
Period: Overall Study
Arm/Group | 1: Venlafaxine Plus Aripiprazole | 2: Placebo Comparator
Started | 91 | 90
Completed | 87 | 83
Not Completed | 4 | 7
Not completed — Adverse Event | 2 | 2
Not completed — subject burden | 2 | 3
Not completed — Lack of Efficacy | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Venlafaxine Plus Aripiprazole | 2: Placebo Comparator | Total
Number analyzed (Participants) | 91 | 90 | 181
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66.4 [62.8 to 71.6] | 65.7 [62.8 to 69.8] | 66.0 [62.8 to 70.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 51 | 103
  Male | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Met Criteria for Remission Based on the Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) is a clinician rated ten item instrument assessing depression symptoms. Possible scores range from 0-60; higher scores indicate greater severity of depression. Remission defined as score of 10 or less based on the MADRS.
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Groups:
- 1: Venlafaxine Plus Aripiprazole; 2: Placebo Comparator: antidepressant (venlafaxine) plus aripiprazol or venlafaxine plus placebo
  venlafaxine XR plus aripiprazole: Dosage of venlafaxine ranged from 150mg to 300mg. Dose of aripirpazole ranged from 2mg to 15mg. Subject remained on venlafaxine throughout the 36 week study. Subject remained on aripiprazole or placebo for up to 24 weeks.
Arm/Group | 1: Venlafaxine Plus Aripiprazole | 2: Placebo Comparator
Number analyzed (Participants) | 91 | 90
percentage of participants | 44 | 29

2. Primary Outcome: Akathisia
Description: Percentage of participants who developed clinically significant akathisia.
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | 1: Venlafaxine Plus Aripiprazole | 2: Placebo Comparator
Number analyzed (Participants) | 91 | 90
percentage of participants | 26.7 | 12.2

3. Primary Outcome: Weight
Description: Weight change in kilograms
Time Frame: Baseline through12 weeks
Population: The number of participants analyzed is lower due to missing data attributable to dropouts. The information obtained is from figure 3B in the manuscript
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | 1: Venlafaxine Plus Aripiprazole | 2: Placebo Comparator
Number analyzed (Participants) | 84 | 85
kilograms | 1.93 (3.00) | 0.01 (3.15)

4. Primary Outcome: Parkinsonism
Description: Percentage of participants who develop signs of parkinsonism
Time Frame: 12weeks
Population: We have a lower number of participants analyzed due to dropouts and missed assessments.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Venlafaxine Plus Aripiprazole | 2: Placebo Comparator
Number analyzed (Participants) | 86 | 81
percentage of participants | 17.4 | 2.5

5. Secondary Outcome: Emergent Suicidal Ideation in Those With no Ideation at the Start of Treatment
Description: percentage of participants who reported suicidal ideation during treatment but not at baseline
Time Frame: 12 weeks
Population: It is a smaller number of participants restricted to those who did not report any suicidal ideation at baseline. This is in Table 3of the manuscript
Measure: Number; unit: percent of participants
Arm/Group | 1: Venlafaxine Plus Aripiprazole | 2: Placebo Comparator
Number analyzed (Participants) | 61 | 65
percent of participants | 21.3 | 29.2

6. Secondary Outcome: QTc Prolongation on EKG (to Greater or Equal to 480 Msec)
Description: percentage of participants
Time Frame: 12 weeks
Population: We had a smaller number of participant observations due to dropouts and missing data. This data is in Table 3 of the manuscript.
Measure: Number; unit: percent of participants
Arm/Group | 1: Venlafaxine Plus Aripiprazole | 2: Placebo Comparator
Number analyzed (Participants) | 78 | 79
percent of participants | 1.3 | 0

ADVERSE EVENTS:
Arm/Group | 1: Venlafaxine Plus Aripiprazole | 2: Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 4/91 | 2/90
Other Adverse Events (participants affected / at risk) | 0/91 | 0/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Venlafaxine Plus Aripiprazole (N=91) | 2: Placebo Comparator (N=90)
completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
hospitalization for MI or CHF (Cardiac disorders) | 1 (1) | 1 (1)
stroke (Nervous system disorders) | 1 (1) | 0 (0)
diverticulitis or excessive vonmiting (Gastrointestinal disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
limited number of participants older than 75, or members of racial/ethnic minority groups; limited follow-up period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No